CLINICAL TRIAL: NCT00408044
Title: Pain After Sternotomy
Brief Title: Dysesthesia Study After Sternotomy
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Mona Momeni, Cliniques Universitaires Saint Luc
Other Study IDs: CE 2005/05SEPT/134
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Ischemic Cardiopathy; Other Forms of Cardiopathy
MeSH Terms: interventions — Cardiac Surgical Procedures; Sternotomy

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: cardiac surgery with sternotomy

SUMMARY:
Chronic pain associated to sternotomy occurs in 40 to 50% of patients after cardiac surgery.

33 to 66% of these patients suffer during 3 month and 25 to 33% have postoperative pain for at least 1 year.

This pain has often negative effects on daily activity. Despite its frequency and importance, the etiology of this chronic pain is not completely understood.

The goal of this study is to understand the mechanism of this chronic pain, to prevent and/or to treat better in the future.

The sensitivity of the thorax after cardiac surgery seems to follow a dynamic evolution which can be observed within several weeks. Therefore we decided to study this evolution.

This study is different from previous ones observing the sensitivity of the thorax at a well defined moment immediately after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with sternotomy

Exclusion Criteria:

* patients with chronic pain
* redo surgery
* patients with neurological pathologies
* patients treated with antidepressant medication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Momeni, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium